CLINICAL TRIAL: NCT03864679
Title: Investigation of Fat and Carbohydrate Oxidation During Moderate Versus Vigorous Intensity Exercise in Healthy Volunteers With Sedentary Lifestyle
Brief Title: Investigation of Fat Oxidation During Moderate Versus Vigorous Intensity Exercise
Acronym: FATOX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Latvian Institute of Organic Synthesis (Other)
Collaborators: Riga East University Hospital (Unknown); University of Latvia (Other); Riga Stradins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Exercise 2018-1
Record Dates: First submitted 2018-06-22; First posted 2019-03-06 (Actual); Last update posted 2019-03-06 (Actual); Status verified 2019-03

CONDITIONS: Healthy; Sedentary Lifestyle
Keywords: exercise; fed; fasted; fat; carbohydrate
MeSH Terms: conditions — Sedentary Behavior; Motor Activity; Lecithin Cholesterol Acyltransferase Deficiency; Platelet Glycoprotein IV Deficiency | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise (Experimental): Subjects will perform a cycling tests
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Subjects will perform a cycling test with 5 min incremental intensity exercise and 1 h cycling test exercising at a moderate-intensity (load will be selected in incremental intensity exercise).

SUMMARY:
Exercise is widely suggested as an important lifestyle change for weight loss, however, the optimal level of intensity moderate versus vigorous remains unclear. It is known that in athletes, during very high-intensity exercise, fat oxidation is decreased and energy is gained mainly from carbohydrate utilization. The aim of this study is to find an optimal workload based on fat oxidation rate during exercise in volunteers with a sedentary lifestyle.

DETAILED DESCRIPTION:
It is planned to recruit 12 healthy volunteers with a sedentary lifestyle in the study group. Since different regimens (fed, fasted and moderate versus vigorous) will be compared in the same subjects, no control group is necessary. Subjects will perform a cycling test with 5 min incremental intensity exercise and 1 h cycling test exercising at a moderate-intensity (load will be selected after the incremental intensity exercise). The expiration of carbon dioxide (CO2) and consumption of oxygen (O2) will be measured, to determine the total fatty acid and carbohydrate oxidation during cycling. Concomitantly, it is planned to measure blood lactate and glucose concentrations during exercise experiments as well as a wide range of blood biochemistry parameters before and after exercise.

The investigators expect to find optimal conditions for the sedentary population for burning of fat, which is the major source of energy during moderate-intensity exercise. Measurements of the fat and carbohydrate oxidation in healthy volunteers with a sedentary lifestyle will contribute to the understanding of exercise regimens for the most effective fat oxidation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Sedentary lifestyle
* BMI 20 - 30 kg/m2
* Be able to attend the laboratory and willing to participate in necessary protocols
* Be willing to undertake the duration of the exercise protocol (3 x 1 hour)
* Have the capacity and willingness to provide informed consent (oral and written)

Exclusion Criteria:

* athletes
* Individuals with chronic cardiovascular disease such as hypertension, valve disease, coronary artery disease, cardiac conduction abnormalities, etc.
* History of pneumothorax or chronic lung disease such as asthma, COPD, bronchiectasis
* Active Smokers
* Pregnant women

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2018-06-18 (Actual); Primary Completion 2018-08-15 (Actual); Study Completion 2018-08-30 (Actual)

PRIMARY OUTCOMES:
Optimal workload | 30 min accelerated load cycling exercise
  The exercise workload (W) for optimal fat burning during exercise
Heart rate change | 30 min accelerated load cycling exercise and 60 min optimal intensity cycling exercise
  Change in heart rate (BPM) from rest to the optimal workload

SECONDARY OUTCOMES:
Influence of fed and fasted state | 30 min accelerated load cycling exercise
  The influence of fed and fasted state on maximal whole body fat oxidation rate during exercise

CONTACTS AND LOCATIONS:
Overall Officials: Ilze Konrade, Principal Investigator — Riga East University Hospital
Locations (1):
- Latvian University, Riga, Latvia

IPD SHARING:
Plan to Share IPD: No